CLINICAL TRIAL: NCT05945641
Title: The Effect of Low-Load Resistance Training Versus High-intensity/Sprint Interval Training on Local Muscle Endurance, Mitochondrial Content, Mitochondrial Function, and Muscle Capillarization
Brief Title: Effect of Low-load Resistance Training vs. High-intensity Interval Training on Local Muscle Endurance
Acronym: LLSIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Cameron Mitchell, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H23-01009
Record Dates: First submitted 2023-06-09; First posted 2023-07-14 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-05

CONDITIONS: Hypertrophy; Muscle Strength; High-Intensity Interval Training; Resistance Training
Keywords: Muscle Strength; Local Muscle Endurance; Muscle Hypertrophy; Mitochondrial Content; Mitochondrial Function; Muscle Capillarization; High-Intensity Interval Training; Sprint Interval Training; Low Load Resistance Training; Resistance Training; Interval Training; Knee Extension; Muscle Endurance
MeSH Terms: conditions — Hypertrophy | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Within subject Design: Each participant will have one leg randomly assigned to each training condition. Training for each leg will occur over the same 12 week training period.
Masking Description: Since the interventions are exercise interventions it is not possible to blind either the participants or Investigator to which condition each participants leg receives. However, the legs will be randomly assigned to their conditions (neither the participant nor the Investigator will determine this.)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low Load Resistance Training (Experimental): LLRET - 12 weeks (2-3 times/week) 3 sets of Knee extension exercise (single leg) done at 30%1- RM. Performed to failure with 3 minutes of rest between sets, weight lifted will be adjusted throughout the study to keep repetitions completed in a 20-30 repetition range.
  Interventions: Behavioral: Low Load Resistance training
- Sprint/High Intensity Interval Training (Experimental): SIT/HIIT- 12 weeks (2-3 times/week), mix of SIT and HIIT (8-15 sets/session). SIT -30 second Super Maximal "Wingate style intervals" performed on a Kicking ergometer (single leg) with 4 minutes rest provided between sets (number of interval ranges from 4-5), load determined from DEXA leg lean mass and will not be altered throughout training.
  HIIT - 1-minute Submaximal efforts (90% single leg kicking ergometer VO2Peak Wattage) performed on a kicking ergometer (single leg) with 1 minute rest provided between sets (number of interval ranges from 8-10), if all sets completed wattage will be increased by 5watts for the next training session.
  Interventions: Behavioral: Sprint/High Intensity Interval Training

INTERVENTIONS:
Behavioral: Low Load Resistance training — Performing single leg knee extension exercise with using equivalent to ~30%1-RM to failure,
  Other Names: LLRET
  Arms: Low Load Resistance Training
Behavioral: Sprint/High Intensity Interval Training — Performing repeated submaximal/maximal 30second-60 seconds (1-3 minute rest between) aerobic intervals on a Kicking ergometer (modified bike that allows cycling to be performed with one leg using a kicking motion).
  Other Names: SIT/HIIT
  Arms: Sprint/High Intensity Interval Training

SUMMARY:
Local muscle endurance (LME) is the ability of a muscle(s) to resist fatigue and is needed for daily activities of life such as climbing stairs, lifting/moving objects, and in sport contexts like rock climbing, mixed martial arts, cross-fit, kayaking and canoeing. Therefore, the investigators want learn how to improve LME and understand what in human bodies changes during exercise training to cause these changes. The investigators know that lifting weights improves muscle strength which is believed to improve LME. Specifically lifting less heavy weights (LLRET) for more repetitions leads to greater gains in LME opposed to heavier weights for fewer repetitions. Therefore, lifting less heavy weights likely causes greater changes in our muscles than lifting heavier weights that cause improvements in LME. Aerobic exercise preformed at high intensities in an interval format (HIIT) may also help improve LME by increasing our muscle's ability to produce energy during exercise. Therefore, the investigators want to see which of LLRET or HIIT leads to greater improvements in LME.

DETAILED DESCRIPTION:
Local muscle endurance (LME) is the ability of a given muscle/muscle group to resist fatigue when performing resistance exercise at a submaximal resistance/load. LME is vital for daily activities of life such as climbing stairs, lifting/moving objects, and in sport contexts such as, rock climbing, mixed martial arts, cross-fit, kayaking and canoeing. Therefore, understanding the mechanisms that underpin LME are of significant interest. Mitochondrial content, mitochondrial function and muscle capillarization have been purported as potential physiological factors that may influence LME. However, currently these mechanisms are speculative in nature and further research is required to draw more conclusive evidence. Furthermore, tolerance to exercise induced discomfort is another a potential mechanism of LME, whereby individuals who train under conditions that induce significant feelings of discomfort may possess a greater capacity to push through discomfort induced via LME tests. However, distinguishing between potential physiological and psychological/neural adaptations regarding LME improvements would require further investigations with nuanced methodology. Low load resistance exercise training (LLRET) has been definitively shown to improve local muscle endurance via numerous investigations. Resistance exercise training (RET), LLRET inclusive improves muscle strength which leads to greater repetition reserve capacity at lower loads. Although, Improvements in muscle strength are not specific to LLRET, yet, LLRET does yield greater gains in LME opposed to high load RET (HLRET). Therefore, LLRET likely induces vital physiological adaptations to greater extent than HLRET that drive improvements in LME such mitochondrial function, mitochondrial content and muscle capillarization. HIIT/Sprint interval training (SIT) induce significant discomfort and improve mitochondrial content/function and muscle capillarization, therefore, HIIT/SIT may be effective interventions to improve muscle endurance.

It is evident that RET of varying loads can improve strength, hypertrophy and LME and that endurance exercise training (EET) improves, VO2 Max, mitochondrial content, mitochondrial function and muscle capillarization. However, minimal research has investigated the impact of RET on single leg maximal aerobic capacity, mitochondrial content, mitochondrial function and muscle capillarization and of EET on muscle strength and muscle hypertrophy and muscle endurance. Furthermore, the findings that do exist from this body of literature are conflicted, with some suggesting RET can improve EET associated adaptions while others suggest no benefit or even decrements in aerobic condition are induced via RET. A similar pattern emerges surrounding the impact of HIIT and SIT on muscle hypertrophy, strength and local muscle endurance, whereby SIT and HIIT may induce gains in hypertrophy, strength and local muscle endurance or may yield no benefit at all. Interestingly, SIT and LLRET fall the closest to one another on the resistance exercise-endurance exercise (RE-EE) continuum suggesting that in theory there would be the largest "crossover" effect from these stimuli. Whereby SIT would elicit the greatest improvements in muscle strength and hypertrophy relative to other EET and LLRET would induce greater enhancement of EET associated adaptations relative to other RET. Although limited research has investigated this potential "crossover effect", evidence suggests that both stimuli may improve single leg maximal aerobic capacity ,mitochondrial content, mitochondrial function, muscle capillarization, muscle strength, muscle hypertrophy and local muscle endurance. However, results are in-consistent between investigations and findings are difficult to compare due to discrepancies in durations of studies, training architecture and intensity of sessions. Furthermore, to date no previous research has directly compared the effect of SIT/HIIT and LLRET on the aforementioned adaptations within the same study, leaving this topic up to speculation. The present study attempts to address this gap in the literature.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and communicate in English
2. 19-30 years of age
3. All "No" answers on the CSEP Get Active questionnaire or doctors' approval to participate
4. Untrained participants: no structured resistance and/or endurance training over the past 12-months (i.e., >2 hours per week of structured/periodized training)

Exclusion Criteria:

1. BMI lower than 18 or greater than 30
2. Current use of cigarettes or other nicotine devices
3. Any major uncontrolled cardiovascular, muscular, metabolic, and/or neurological disorders
4. Any medical condition impacting the ability to participate in maximal exercise
5. Type one or type two diabetes
6. Diagnosis of cancer or undergoing cancer treatment in the past 12 months
7. Taking blood-thinning medication or the presence of a bleeding disorder
8. Drug therapy with any drugs that alter skeletal muscle metabolism (i.e., Metformin, Benzodiazepines)

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-27 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Change in repetitions completed for 30% pre-training 1- Repetition maximum (Single leg Knee extension) | Change from baseline to 6 weeks
  The number of single leg knee extension repetitions that one can complete at 30% of their pre-training 1-RM
Change in Repetitions completed for 30% pre-training 1- Repetition maximum (Single leg Knee extension) | Change from baseline to 12 weeks
  The number of single leg knee extension repetitions that one can complete at 30% of their pre-training 1-RM
Change in CFPE index (Capillary to fiber ratio normalized to fiber perimeter) | Change from baseline to 12 weeks
  Mean number of capillaries touching each muscle fibre (normalized to the fibre perimeter). Assessed using imaging of muscle samples gathered via muscle biopsies.
Change in Maximal Citrate synthase (CS) Activity | Change from baseline to 12 weeks
  Indicator of Mitochondrial content and function in skeletal muscle.

SECONDARY OUTCOMES:
Change in Single leg Knee extension 1- Repetition maximum (weight lifted) | Change from baseline to 6 weeks
  Maximum Weight lifted for 1 repetition of single leg knee extension exercise.
Change in Single leg Knee extension 1- Repetition maximum (weight lifted) | Change from baseline to 12 weeks
  Maximum Weight lifted for 1 repetition of single leg knee extension exercise.
Change in Single leg Knee extension Isometric Maximum Voluntary Contraction | Change from baseline to 6 weeks
  Maximal force production at 90 degrees of knee flexion. Assessed via Biodex
Change in Single leg Knee extension Isometric Maximum Voluntary Contraction | Change from baseline to 12 weeks
  Maximal force production at 90 degrees of knee flexion. Assessed via Biodex
Change in Single leg Knee Flexion Isometric Maximum Voluntary Contraction | Change from baseline to 6 weeks
  Maximal force production at 90 degrees of knee flexion. Assessed via Biodex
Change in Single leg Knee Flexion Isometric Maximum Voluntary Contraction | Change from baseline to 12 weeks
  Maximal force production at 90 degrees of knee flexion. Assessed via Biodex
Change in Single leg Knee Flexion Isokentic Maximum Voluntary Contraction | Change from baseline to 6 weeks
  Maximal force production at 60 degrees/second. Assessed via Biodex
Change in Single leg Knee Flexion Isokentic Maximum Voluntary Contraction | Change from baseline to 12 weeks
  Maximal force production at 60 degrees/second. Assessed via Biodex
Change in Single leg Knee Extension Isokentic Maximum Voluntary Contraction | Change from baseline to 6 weeks
  Maximal force production at 60 degrees/second. Assessed via Biodex
Change in Single leg Knee Extension Isokentic Maximum Voluntary Contraction | Change from baseline to 12 weeks.
  Maximal force production at 60 degrees/second. Assessed via Biodex
Change in Single leg VO2 Peak on Kicking ergometer (ml/kg leg lean mass/min) | Change from baseline to 12 weeks.
  Maximal Oxygen consumption/minute of single leg.
Change in Single leg Wingate test on kicking ergometer (Max Power) | Change from baseline to 6 weeks
  maximum 5 second power achieved during Single leg Wingate test on kicking. ergometer
Change in Single leg Wingate test on kicking ergometer (Max Power) | Change from baseline to 12 weeks
  maximum 5 second power achieved during Single leg Wingate test on kicking. ergometer
Change in Leg lean mass | Change from baseline to 12 weeks.
  Assessed via Dual X-ray absorptiometry. Measured in Kg.
Change in Vastus Lateralis Cross sectional area (CSA) | Change from baseline to 12 weeks.
  CSA of vests laterals muscle assessed via ultrasonography.
Change in Type I and II Fiber Cross sectional area (CSA) | Change from baseline to 12 weeks
  Mean CSA of Type I and II muscle fibers using imaging of muscle samples gathered via muscle biopsies.
Change in Capillary to fiber ratio (C/FI) | Change from baseline to 12 weeks
  Mean number of capillaries touching each muscle fibre. Assessed using imaging of muscle samples gathered via muscle biopsies.

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy if British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be held by Lucas Wiens and will be released upon request to other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be made available after publication/completion of the project. Data will remain available for at least 10 years following the completion of this project.
Access Criteria: Data will only be released to researchers who have valid association with an institution or private laboratory.